CLINICAL TRIAL: NCT01561937
Title: Use of Recombinant FVIIa to Mitigate Warfarin Anticoagulation Therapy-Mediated Bleeding in a Single Centre, Randomized, Placebo-controlled, Double-blind Clinical Trial
Brief Title: Use of Activated Recombinant Human Factor VII to Reduce Bleeding Caused by Warfarin Treatment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: F7HAEM-1825
Record Dates: First submitted 2012-03-21; First posted 2012-03-23 (Estimated); Last update posted 2016-11-25 (Estimated); Status verified 2016-11

CONDITIONS: Haemostasis; Healthy
MeSH Terms: interventions — Warfarin; Factor VII

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pre-warfarin treatment (trial part A) (Experimental)
  Interventions: Drug: warfarin
- Post-warfarin treatment (trial part B) (Experimental)
  Interventions: Drug: eptacog alfa (activated); Drug: placebo

INTERVENTIONS:
Drug: warfarin — After a baseline punch biopsy (B0), warfarin is administered over a period of approximately 7-14 days. Dose is adjusted individually to achieve INR target. Once a stable INR is achieved, a second biopsy (B1) will be performed
  Arms: Pre-warfarin treatment (trial part A)
Drug: eptacog alfa (activated) — If the subject is eligible to continue in trial part B, trial drug will be administered i.v. as a slow bolus injection over 2 to 5 minutes in five different doses followed by two biopsies (B2) and (B3) 15 minutes and 5 hours and 15 minutes, respectively, after trial drug administration
  Other Names: activated recombinant human factor VII
  Arms: Post-warfarin treatment (trial part B)
Drug: placebo — If the subject is eligible to continue in trial part B, trial drug will be administered i.v. as a slow bolus injection over 2 to 5 minutes in five different doses followed by two biopsies (B2) and (B3) 15 minutes and 5 hours and 15 minutes, respectively, after trial drug administration
  Arms: Post-warfarin treatment (trial part B)

SUMMARY:
This trial is conducted in the United States of America (USA). The aim of this trial is to evaluate the efficacy of activated recombinant human factor VII to mitigate experimentally-induced bleeding in healthy volunteers treated with warfarin to reach a targeted INR (International Normalization Ratio).

ELIGIBILITY:
Inclusion Criteria:

* INR below or equal to 1.2

Exclusion Criteria:

* The receipt of any investigational drug within 1 month prior to this trial
* Use of anticoagulation therapy-defined as vitamin K antagonists, platelet antagonists, heparin (or low molecular weight heparin), aspirin or NSAIDs (Non-Steroidal Anti-Inflammatory Drug) within 14 days prior to trial
* African-American race
* Weight above 160 kg
* Supplemental Vitamin K use

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2007-01; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Bleeding duration measured in minutes after biopsies in trial part A | From onset of bleeding till the end of the bleeding
Bleeding duration measured in minutes after biopsy B1 in trial part B | From onset of bleeding till the end of the bleeding

SECONDARY OUTCOMES:
Blood volume reported in millilitres after biopsies in trial part A | From onset of bleeding till the end of the bleeding
Blood volume reported in millilitres after biopsy B1 in trial part B | From onset of bleeding till the end of the bleeding
Adverse events, including thrombotic events | From day 0 to days 14-28
Change in coagulation-related parameters after biopsy B1 | From baseline to 3 hours after B1
Change in coagulation-related parameters after biopsy B2 | From baseline to 3 hours after B2
Change in coagulation-related parameters after biopsy B3 | From baseline to 3 hours after B3
Clot dynamics: R in minutes (trial part B) | Time to onset of clot formation
Clot dynamics: K in minutes (trial part B) | Time to achieve 20mm clot strength

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Overland Park, Kansas, United States

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com